CLINICAL TRIAL: NCT06604741
Title: Comparison of High Volume Intensity Training and Low Volume Intensity Training With IMT on Pulmonary Function and Breathing Efficiency of Recreational Swimmers
Brief Title: High vs Low Volume Intensity Training With IMT On Pulmonary Function And Breathing Efficiency On Recreational Swimmers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Sumayya Karim
Record Dates: First submitted 2024-09-18; First posted 2024-09-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy Young Adults
Keywords: Inspiratory muscle training; High volume intensity training; Low volume intensity training; Swimmers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High volume intensity (HVIMT) (Experimental): High-volume intensity inspiratory muscle training (IMT) is a therapeutic approach designed to improve respiratory muscle strength and endurance. In this clinical trial, participants will engage in a structured regimen of inspiratory exercises with high resistance and significant repetition volume.
  Participants will perform inspiratory muscle exercises using power breath that provides high resistance, with a focus on both intensity and volume. The protocol involves 3 sessions per day for 6 weeks.
  Interventions: Other: Assigned interventions for HVIMT
- Low volume intensity LVIMT (Experimental): Participants will engage in a structured training program involving inspiratory muscle exercises with high resistance and a high volume of repetitions. The regimen includes multiple sessions per day over several weeks, using specialized inspiratory muscle training devices.
  Changes in inspiratory muscle strength (measured by maximal inspiratory pressure) and endurance.
  Interventions: Other: Assigned Interventions for LVIMT

INTERVENTIONS:
Other: Assigned Interventions for LVIMT — IMT is a form of exercise designed to strengthen the muscle involved inhalation, primarily the diaphragm and intercostal muscles.
  The LVIMT group will perform IMT once daily, 5 days a week, maintaining 60% of maximal inspiratory pressure (MIP) throughout the 6-week intervention.
  The intervals are typically longer in duration (e.g., 2-4 minutes) with a work-to-rest ratio of 1:1 or 1:0.5.
  POSITION: rested and seated position. FREQUENCY: more frequency, once a day. 2-3 sessions per week. INTENSITY: Low resistance. Only 60%% MIP. TIME: shorter duration of 10-20 mint.
  Arms: Low volume intensity LVIMT
Other: Assigned interventions for HVIMT — The HVIMT group is trained twice daily, with the morning session matching the LV-IMT protocol, and an additional afternoon session. The HVIMT group also experienced a progressive increase in intensity, starting at 60% MIP and reaching 80% by the end of the study. LVIMT works for beginner or individuals with limited respiratory capacity while HVIMT is used for individual with high baseline respiratory fitness.
  The intervals are typically shorter in duration (e.g., 30 seconds to 2 minutes) with a work-to-rest ratio of 1:1 or 1:2.
  POSITION; Seated upright position. FREQUENCY: more frequency two session per week. 4-5 sessions per week. INTENSITY: high resistance. 60%-80% MIP.
  (gradual increment the load by 10% every 2 weeks to reach 80% MIP)
  TIME: longer duration 20-30 mint.
  Arms: High volume intensity (HVIMT)

SUMMARY:
This study aims to evaluate the impact of inspiratory muscle training (IMT) on respiratory function and swimming performance in competitive swimmers. Given the importance of optimal respiratory function in swimming, this trial investigates whether IMT can improve swimming performance metrics, such as lap times and endurance, and overall respiratory health.

DETAILED DESCRIPTION:
Effective respiratory function is crucial for swimmers, given the demanding nature of the sport. Inspiratory muscle training (IMT) has been shown to improve respiratory muscle strength and endurance in various populations. This study aims to explore the effects of IMT specifically on competitive swimmers, assessing both physiological and performance-related outcomes. To assess whether a structured IMT program improves swimming performance, respiratory muscle strength, and overall respiratory efficiency in recreational swimmers. A randomized controlled trial involving 56 competitive swimmers will be conducted. The study duration will be 8 weeks, with assessments conducted at baseline, mid-point, and at the end of the intervention. The IMT groups will participate in a 20-30 minute training session, 4 to 5 times per week, using power breath device . The training will focus on enhancing inspiratory muscle strength and endurance. This study aims to provide robust evidence on the benefits of IMT for swimmers, potentially informing future training practices and enhancing competitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female Swimmers
* Age; 18-25
* Minimum of 2 years of regular swimming training experience, with at least 3 swimming sessions per week.

Exclusion Criteria:

* Refusal to participate in the study.
* History of respiratory or cardiovascular conditions that could impact participation or results.
* Participation in any other respiratory or exercise-related intervention study within the last 6 months.
* Consumption of any medications or supplements that could potentially influence respiratory or cardiovascular function.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Peak Expiratory Flow Rate (PEFR) | 6 weeks
  Peak expiratory flow rate (PEFR) Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
Forced Vital Capacity (FVC) | 6 weeks
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
  Changes in FVC from baseline to 3rd week and after 6 weeks day of intervention will be assessed.
Forced Expiratory volume in 1sec (FEV1) | 6 weeks
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
Swimming efficiency (SWOLF) score | 6 weeks
  A SWOLF score is a metric used in swimming to assess efficiency. It combines the time it takes to swim a distance (in seconds) with the number of strokes taken to complete that distance.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD, Principal Investigator — Riphah International University
Locations (1):
- Bahira Active Club., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No